CLINICAL TRIAL: NCT06772675
Title: Implementing Vancomycin Reducing Practices (VRP) in Preterm Infants
Brief Title: Vancomycin Reduction Practices (VRP) in the NICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sagori Mukhopadhyay, Principal Investigator, Attending Neonatologist, Associate Professor of Pediatrics, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-021976; GRT-00003877 (Other Grant/Funding Number: Agency for Health Care Research and Quality)
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-06

CONDITIONS: Antibiotic Stewardship; Neonatal Sepsis, Late-Onset; Vancomycin
Keywords: implementation study
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: Cluster randomized study of external facilitation as an implementation strategy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sites receiving external facilitation (Experimental): Sites will receive guidance from an external facilitator to support uptake of the VRP.
  Interventions: Behavioral: External Facilitation
- Sites not receiving external facilitation (No Intervention): Sites will not receive guidance from an external facilitator.

INTERVENTIONS:
Behavioral: External Facilitation — Designated external facilitators will conduct monthly meetings with local champions at each site. Designated facilitators will follow the developed facilitation guide, that includes content area to cover in each meeting, case scenarios as examples, and tips on how to communicate and support the internal facilitators. The goal is to enable problem-solving and support the local champion in implementing VRP with fidelity
  Arms: Sites receiving external facilitation

SUMMARY:
This multi-center, cluster randomized study aimed at improving implementation of vancomycin reducing practices (VRP) in neonatal intensive care units (NICUs). Sites will be recruited and randomized to receive either external facilitation or no external facilitation to assess the effect on center-level fidelity to the core components of VRP implementation. Interventions available to both study arms are directed at hospital staff and includes identification of local champions, educational outreach, unit-level audit & feedback, and use of a clinical decision support tool.

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU
* Affiliated with Kaiser Permanente Northern California (KPNC) or Children's Hospital of Philadelphia Newborn Care Network (CNBCN)
* Recruited by study team

Exclusion Criteria:

* Site not recruited for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Fidelity of VRP use | 2.5 years - From beginning of implementation phase to the end of the sustainment phase
  Proportion of late onset sepsis (LOS) evaluations performed with high fidelity. High fidelity is defined when the evaluation follows all three core components of VRP use.

SECONDARY OUTCOMES:
Appropriateness/acceptability | 2.5 years - From beginning of implementation phase to the end of the sustainment phase
  Response to questions about whether vancomycin reducing practices (VRP) was agreeable and/or a good fit for the unit measured using validated instruments comprising of 5-point Likert scales (Weiner et al). Participants are offered options ranging from completely disagree (1) to completely agree (5), with higher scores indicating a higher degree of acceptability or feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Sagori Mukhopadhyay, MD, MMSc, Principal Investigator — Children's Hospital of Philadelphia
Locations (13):
- United States (13):
  - Kaiser Permanente Modesto Medical Center, Modesto, California
  - Kaiser Permanente East Bay - Oakland Medical Center, Oakland, California
  - Kaiser Permanente Roseville Medical Center, Roseville, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - Kaiser Permanente San Leandro Medical Center, San Leandro, California
  - Kaiser Permanente Santa Clara Medical Center, Santa Clara, California
  - Kaiser Permanente Walnut Creek Medical Center, Walnut Creek, California
  - Medical Center of Princeton, Plainsboro, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
Participants here are the clinicians at the sites randomized to external facilitation. The investigators obtain survey (de-identified) and interview data from representative group of the clinicians. Since the investigators will be gathering richly detailed qualitative data that, even if de-identified of names or locations, can still be linked back to sites or individuals, the investigators will not share interview data for secondary analysis or use beyond the purposes of the proposal. The investigators will maintain de-identified (for both site and respondent identifiers) survey output that can be shared upon appropriate request to the principal investigator.